CLINICAL TRIAL: NCT06635031
Title: Assessment of the Relationship Between Sense of Coherence and the Healing of Surgery-related Intraoral Wound by Using a Novel Scale: A Clinical Randomized Study.
Brief Title: The Relationship Between Sense of Coherence and Wound Healing.
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: 23/77
Record Dates: First submitted 2024-09-24; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-11

CONDITIONS: Wound Heal; Sense of Coherence
MeSH Terms: interventions — Surgery, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Oral surgery — The patients were undergone routine oral surgeries. Surgical procedures included an incision on the oral mucosa and full-thickness flap reflection, and the primary wound closure was achieved by polyglactin absorbable sutures.

SUMMARY:
The study aimed to investigate the relationship between sence of coherence (SOC) and surgery-related oral wound healing.

The study was consisted of one hundred and sixty patients of both sexes (female,male) who were scheduled for oral surgery. Pre-operatively the patients were asked to complete a questionnaire designed to measure their Sense of Coherence (SOC). The wound healing was evaluated after 4 days, 14 days and 6 weeks after surgical operation. The results were analyzed statistically.

DETAILED DESCRIPTION:
Many factors play a role in wound healing (WH) including physiologic factors. The concept of Sense of Coherence (SOC), reflects an individual's capacity to respond to stressful situations. High SOC scores indicate a strong SOC, and individuals with strong SOC are reported to tolerate stress better. Additionally, a strong SOC has been associated with fewer symptoms and significantly fewer issues related to oral condition. The aim of this study is to evaluate the relationship between SOC and wound healing following oral surgery. The study included 160 patients of both sexes (female,male). An informed consent form was obtained from all participants. Pre-operatively the patients were asked to complete a questionnaire designed to measure their Sense of Coherence (SOC). A blinded operator, who was not involved in the operation, recorded all data of the patients pre-operatively. All patients were undergone oral surgery. All surgical procedures were performed by the second maxillofacial surgeon. The first blinded operatoand conducted postoperative measurements. The wound healing was evaluated after 4 days, 14 days and 6 weeks after surgical operation. To evaluate of wound healing, a scale named Inflammatory Proliferative Remodeling (IPR) Scale was used. According to this scale, patients were recalled 3 days, 14 days and 6 weeks after surgical operation. The third blinded researcher was responsible for the analysis data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18-65 years
* Patients classified as American Society of Anesthesiologists (ASA) physical status ASA I
* Patients scheduled to undergo oral surgery

Exclusion Criteria:

* Not consenting to participate
* Intake of steroid, bisphosphonate or immune-suppressive medication
* Receiving radiotherapy in the head and neck area
* Pregnancy
* Inability to self-evaluate, and inability to communicate verbally and in writing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred and sixty adult patients of both sexes
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Sence of Coherence | 6 weeks
  Sence of Coherence (SOC) was measured using a 13-question survey, where participants rate their answers on a scale from 1 to 7, with 1 representing "never" and 7 indicating "very often." Total scores above 45 are regarded as indicative of high SOC values.
Evaluation of Oral Wound Healing | 6 weeks
  Wound Healing (WH) was assessed by using a scale called Inflammatory Proliferative Remodeling (IPR) Scale. According to the scale, each phase of the healing is scored based on the parameters, including edema, bleeding, swelling. The total score of the IPR scale ranges from 0 to 16; 0-4 indicates poor healing; 5-10, acceptable healing; and 11-16, excellent healing.

SECONDARY OUTCOMES:
Evaluation of post-operative pain | 6 weeks
  To measure pain, participants were asked to describe their pain at follow-up appointments using a Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain.
  The numerical values obtained from these two scales were subjected to statistical analysis, to determine if there was a relationship between Sence of Coherence and post-operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: ALANUR ÇİFTÇİ ŞİŞMAN, PhD, DDS, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)